CLINICAL TRIAL: NCT05767411
Title: The Effect of Asymmetric Postural Loading on the Movement of the Right Hemidiaphragm
Brief Title: Asymmetric Movement of the Diaphragm
Status: Completed | Type: Observational
Sponsor: University Hospital, Motol (Other)
Responsible Party: Principal Investigator, Martin Sembera, Clinical Professor, University Hospital, Motol
Other Study IDs: EK-224/23
Record Dates: First submitted 2023-03-02; First posted 2023-03-14 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to investigate the movement of the right hemidiaphragm when lifting a load with the left and right hand.

DETAILED DESCRIPTION:
Hemidiaphragm movement will be assessed by m-mode ultrasonography in a standing position. The study will include 30-40 healthy adult volunteers. The examination will consist of two tidal inspirations and expirations, two inspirations and expirations during lifting the kettlebell with the left hand and two inspirations and expirations during lifting the kettlebell with the right hand. The weight of the kettlebell will correspond to about 10% of the participant's body weight.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Able to comply with the study protocol, in the investigator's judgment
* Aged 18-40 years, inclusive
* Healthy as determined by the Investigator based on medical history, physical examination, vital signs and neurological examination
* Waist-to-height ratio < 0,59

Exclusion Criteria:

* Low back pain (acute or chronic)
* Previous abdominal or spine surgery
* Acute or chronic respiratory or musculoskeletal disorder
* Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks before initiation of the study
* Pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy Subjects
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-06-14 (Actual); Study Completion 2023-06-21 (Actual)

PRIMARY OUTCOMES:
Hemidiaphragm movement | 7 months
  Distance of the diaphragm from the ultrasound transducer in millimeters during tidal breathing, and when lifting a load with the left and right hand.

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Kolar, Prof, PhD, Study Chair — Department of Rehabilitation and Sports Medicine, University Hospital Motol, Prague, Czech Republic
Locations (1):
- Pavel Kolar´s Centre of Physical Medicine, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Undecided